CLINICAL TRIAL: NCT01681706
Title: HIV Indicator Diseases Across Europe Study
Acronym: HIDES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jesper Grarup (Other)
Responsible Party: Sponsor-Investigator, Jesper Grarup, Director of Administration, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: HIDES
Record Dates: First submitted 2012-08-28; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: HIV
Keywords: HIV; Indicator disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this non-interventional study is to implement a survey initiative to assess HIV prevalence for one or more diseases and/or conditions within a specific segment of the population not yet diagnosed with HIV, who presents for care with the specific disease/condition.

The list of diseases below is not indicative of the most important indicator diseases for HIV but rather a list of diseases suggested for surveillance.

This study will enrol patients presenting with the following diseases/conditions:

1. Presenting for care of malignant lymphoma, irrespective of type
2. Presenting for care of cervical or anal dysplasia or cancer, (Cervical CIN II and above)
3. Presenting for care of Hepatitis B or C virus infection (acute or chronic - and irrespective of time of diagnosis relative to time of survey),
4. Presenting with ongoing mononucleosis-like illness
5. Presenting with unexplained leukocytopenia or thrombocytopenia lasting at least 4 weeks
6. Presenting with seborrheic dermatitis / exanthema
7. Presenting with pneumonia, admitted to hospital for at least 24h
8. Presenting with unexplained lymphadenopathy
9. Presenting with peripheral neuropathy of unknown cause (diagnosed by neurologist)
10. Presenting with primary lung cancer
11. Presenting with severe or recalcitrant psoriasis (newly diagnosed)

DETAILED DESCRIPTION:
Most patients infected with HIV across the European continent remain undiagnosed; although this percentage varies markedly from 15-80% across the continent. Undiagnosed HIV is harmful to the person infected as appropriate health interventions are then delayed until the HIV infection is diagnosed. It is also detrimental to society as persons unaware of their HIV infection may transmit more frequently to others than persons that are aware of their HIV status.

An important public health issue is hence how to diagnose more HIV-infected persons earlier in the course of their infection. In the US, the Centers for Disease Control and Prevention (CDC) has introduced testing guidelines where all persons are tested upon entry into the hospital system (the "opt-out" testing guidelines).

At the "HIV in Europe" conference held in November 2007, the general sense was that such an approach would not be suitable for Europe. Conversely, the conference recommended further development of focused HIV testing in patients presenting with certain clinical conditions and/or diseases (i.e. indicator condition guided testing).

Cost effectiveness analyses suggests cost savings if a population with a HIV prevalence of 1% or more are tested although this rate may be as low as 0.1%. However, there is very little - if any - evidence on HIV prevalence for various conditions and diseases in specific and easy to identify sections of society. This is true in general and particularly across the European continent.

Surveys will be undertaken by the investigators:

Zangerle, Kitchen, U H Innsbruck, Vassilenko, Minsk Municipal Infectious Diseases Hospital, Necsoi, Clumeck, Saint-Pierre U H Hadziosmanovic, U of Sarajevo Begovac, U Hospital of Infectious Diseases Pedersen, Mogensen, Abildgaard, Titlestad, Odense U H Dragsted, Roskilde H Späth, U of Bonn Sthoeger, Neve-Or AIDS Centre d'Armino Monforte, Mareo, Comi, Centanni, San Paolo H Grzeszczuk, Medical U of Bialystok Maltez, H Curry Cabral Castro, HU A Coruna-Hospital Juan Canalejo Masia, HU Elche Estrada, HCU San Carlos Iribarren, H. Donostia Ortega, CH General de Valencia Ocampo, H Xeral-Cies Vernazza, Kantonsspital St. Gallen Perry, Fisher, Elton John Centre, Morris, RIDU Minton, St James's U H Palfreeman, Leicester Royal Infirmary Gazzard, Sullivan, ChelseaWestminster H Winston, Walsh, St Mary's H Anderson, Millett, Homerton H NHS Trust Farazmand, Huddersfield Royal Infirmary Ong, Krasnov, Kharkov Regional Clinic of Infectious Diseases Kutsyna, State Medical U

ELIGIBILITY:
Inclusion Criteria:

* HIV status unknown
* Presenting for care with 1 of the 11 indicator diseases surveyed.

Exclusion Criteria:

* Known HIV positive

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants between the age of 18 and 64 years old, presenting with 1 of the 11 indicator diseases surveyed
Sampling Method: Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HIV | Participants are surveyed once up to month 23 for presenting indicator disease and result of the HIV test performed. Per site 100 participants are included in each survey - in total the single survey requires minimum 400 participants from all sites
  To assess the HIV prevalence for the identified diseases and/or conditions within a specific segment of the population not yet diagnosed with HIV and that present for care with the specific disease/condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Lundgren, Prof., Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Panum Institute, Health faculty,, Copenhagen, Copenhagen, Denmark